CLINICAL TRIAL: NCT07048366
Title: Art as a Therapeutic Tool in the Rehabilitation of Patients With Fibromyalgia: the University Museum as a Setting for an Integrative Medicine Program - a Randomized Controlled Trial
Brief Title: Mindfulness-based Rehabilitation in a University Museum Setting to Reduce Pain and Improve Quality of Life in Women With Fibromyalgia: a Randomized Controlled Trial
Acronym: FMmuseo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Teresa Paolucci, Associate Professor, MD, PhD, Physical and Rehabilitation Medicine, G. d'Annunzio University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 401144/25
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Fibromyalgia; Chronic Pain; Musculoskeletal Pain
Keywords: Fibromyalgia; Rehabilitation; Integrative Medicine; Art Therapy; Museums
MeSH Terms: conditions — Fibromyalgia; Chronic Pain; Musculoskeletal Pain | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: Participants with fibromyalgia will be randomly assigned in a 1:1 ratio to either the integrated rehabilitation program conducted in the museum setting or to a control group receiving the same mindfulness-based intervention at the CARES (Center for Disability, Rehabilitation and Sports Medicine), at University . Both groups will be followed in parallel for the study duration.
Who Masked: Participant, Outcomes Assessor
Masking Description: This study employs a double-blind design where both participants and outcome assessors are masked to the intervention assignment. Participants are unaware of their group allocation (treatment vs. control). Personnel collecting and analyzing outcome data will also be blinded to group assignment to minimize bias. The care providers delivering the intervention, due to the nature of the behavioral therapy, may not be fully masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Museum-Based Integrated Rehabilitation Group (Experimental): Participants in this arm will receive an 8-week integrated rehabilitation program conducted at the University Museum. The program consists of weekly 60-minute sessions that incorporate mindfulness techniques, conscious breathing exercises, body scan meditation, mindfulness walking within the museum's exhibition spaces, specific stretching and mobilization techniques, and gratitude and recognition exercises, all framed by the artistic and cultural context of the museum.
  Interventions: Behavioral: Integrated Rehabilitation Program at the University Museum
- CARES Control Group (Active Comparator): Participants in this arm will receive the same mindfulness-based integrated rehabilitation program delivered at the CARES (Center for Disability, Rehabilitation and Sports Medicine), at University. This group will serve as the control arm for comparison with the experimental museum-based intervention.
  Interventions: Other: CARES treatment

INTERVENTIONS:
Behavioral: Integrated Rehabilitation Program at the University Museum — This intervention consists of an 8-week integrated rehabilitation program, with weekly 60-minute sessions, conducted at the University Museum. The program includes mindfulness techniques, conscious breathing exercises, body scan meditation, mindfulness walking within the museum's exhibition spaces, specific stretching and mobilization techniques, and gratitude and recognition exercises, all framed by the artistic and cultural context of the museum. The museum environment is utilized as a therapeutic setting to amplify the benefits of the behavioral techniques.
  Arms: Museum-Based Integrated Rehabilitation Group
Other: CARES treatment — Participants in the control arm will receive the same mindfulness-based integrated rehabilitation program delivered at the CARES University Center. The intervention consists of eight weekly 60-minute sessions including breathing awareness, body scan, mindful walking, and guided mindfulness exercises. This program mirrors the structure and duration of the museum-based intervention but takes place in a conventional rehabilitation setting.
  Arms: CARES Control Group

SUMMARY:
This research study aims to investigate whether art and integrative medicine, within a unique setting like a university museum, can offer a new approach to help women suffering from fibromyalgia. Fibromyalgia is a chronic condition causing widespread pain and other symptoms such as fatigue and sleep disturbances. The question this study seeks to answer is: Is an 8-week rehabilitation program, based on mindfulness and body awareness techniques, conducted at the University Museum of the G. d'Annunzio University, effective in reducing pain and improving the quality of life (physical and mental well-being) and coping abilities in female fibromyalgia patients? Participants will be randomly assigned to either receive this program in the museum or to a control group.

DETAILED DESCRIPTION:
Fibromyalgia Syndrome (FM) is a complex and debilitating chronic musculoskeletal pain condition characterized by widespread pain, tenderness, and a myriad of associated symptoms including profound fatigue, sleep disturbances, cognitive impairment (often referred to as "fibro-fog"), and affective disorders such as anxiety and depression. Its prevalence is significant, affecting a substantial portion of the global population, predominantly women. Diagnosis relies on established criteria (e.g., ACR 1990, revised 2010/2011, and 2016 criteria), emphasizing the presence of widespread pain and symptom severity. The underlying pathophysiology is multifactorial, involving neuro-immuno-endocrine dysregulation, central sensitization (an amplification of pain signals in the central nervous system), and in some cases, small fiber neuropathy, leading to an altered pain perception.

Given its complex nature, a purely pharmacological approach to fibromyalgia is often insufficient. Current evidence strongly supports a multifactorial therapeutic strategy that integrates pharmacological treatments with non-pharmacological interventions, including complementary therapies and integrated medicine. This study introduces a novel, non-pharmacological integrated rehabilitation pathway designed to address the multifaceted symptoms of fibromyalgia.

This randomized controlled trial investigates the efficacy of a unique integrated rehabilitation program delivered within the evocative environment of a university museum. The program leverages the principles of art therapy and neuroaesthetics, combined with established mindfulness and body awareness techniques, to create a holistic and immersive healing experience. The rationale is rooted in the understanding that engagement with art and culturally enriching environments can positively influence brain function and emotional states. Specifically, interactions within a museum setting are hypothesized to:

* Stimulate the brain's reward system, fostering positive emotions and reducing pain perception.
* Modulate cortical maps, potentially normalizing altered somatosensory processing observed in fibromyalgia.
* Provide a powerful distraction from chronic pain and discomfort, shifting focus towards aesthetic appreciation and inner experiences.
* Enhance emotional regulation and promote self-efficacy in managing symptoms.
* The museum itself acts as a "setting of care," providing a calming and inspiring atmosphere that can amplify the therapeutic effects of rehabilitation, reducing stress and promoting overall well-being.

The intervention consists of an 8-week program with weekly 60-minute sessions. Participants in the experimental group engage in a structured curriculum that integrates various techniques, including conscious breathing exercises, body scan meditation, mindfulness walking within the museum's exhibition spaces, specific stretching and mobilization techniques, and gratitude and recognition exercises, all framed by the artistic and cultural context of the university museum. This approach aims to cultivate body awareness, reduce pain catastrophizing, and improve emotional coping mechanisms.

Participants with a confirmed diagnosis of fibromyalgia will be randomly assigned (1:1 ratio) to either this museum-based integrated therapy group or a control group (e.g., a waitlist for conventional treatments). The study is designed to rigorously evaluate the impact of this innovative approach on primary and secondary outcome measures, including pain reduction, improvement in quality of life, and enhanced coping strategies. Ethical considerations, including informed consent and participant safety, are paramount, and the study adheres to the principles of the Declaration of Helsinki. The sample size has been determined through a power calculation to ensure statistical validity, aiming to detect a clinically significant reduction in pain as the primary outcome.

This study seeks to provide robust evidence for the therapeutic potential of art and integrated medicine in the management of fibromyalgia, potentially offering a valuable, accessible, and non-pharmacological addition to existing treatment paradigms.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Diagnosis of Fibromyalgia Syndrome according to 2016 criteria
* Muscle pain Visual Analogue Scale (VAS) score greater than 5 in the last month
* Age between 18 and 60 years
* Absence of other chronic, widespread, or localized painful conditions
* Absence of any other condition that might affect pain perception (e.g., diabetes)
* Absence of neurological or psychiatric conditions that might affect study participation
* Absence of current or past oncological diseases in the last 5 years
* Absence of corticosteroid therapy in the last 30 days
* Absence of NSAID (Non-Steroidal Anti-Inflammatory Drugs) and analgesic therapy in the last 4 days
* Absence of pregnancy and breastfeeding for the entire duration of observation
* Signed informed consent

Exclusion Criteria:

* Presence of severe scoliosis or kyphoscoliosis
* Previous spinal surgeries or sequelae of vertebral fractures
* Presence of lumbosciatalgia (sciatica-like pain in the lower back) at the time of the visit
* Presence of osteoporosis
* Presence of neurological or psychiatric conditions
* Current therapy with corticosteroids and/or NSAIDs and/or analgesics
* Pregnancy or breastfeeding

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only female participants with a diagnosis of Fibromyalgia Syndrome are eligible to participate.
Enrollment: 44 (Estimated)
Dates: Start 2025-11-27 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Pain Reduction | Baseline (T0), End of treatment (T1, after 8 weeks), Follow-up (T2, 4 weeks after end of treatment).
  Reduction in musculoskeletal pain intensity, evaluated by Visual Analogue Scale (VAS) for musculoskeletal pain (0-10 cm score).

SECONDARY OUTCOMES:
Quality of Life Improvement | Baseline (T0), End of treatment (T1, after 8 weeks), Follow-up (T2, 4 weeks after end of treatment).
  Improvement in the physical and mental dimensions of quality of life. Metric: SF-12 (Short Form-12 Health Survey) total score (0-100).
Fibromyalgia Impact on Daily Life | Baseline (T0), End of treatment (T1, after 8 weeks), Follow-up (T2, 4 weeks after end of treatment).
  Changes in the impact of fibromyalgia on daily activities and overall functioning. Metric: Fibromyalgia Impact Questionnaire (FIQ) scores (ranging from 0 to approximately 100).
Global Symptom Severity | Baseline (T0), End of treatment (T1, after 8 weeks), Follow-up (T2, 4 weeks after end of treatment).
  Changes in the overall severity of symptoms associated with fibromyalgia. Metric: Fibromyalgia Status Scale (FSS) scores (0-10 for each item).
Anxiety Levels | Baseline (T0), End of treatment (T1, after 8 weeks), Follow-up (T2, 4 weeks after end of treatment).
  Changes in anxiety symptoms. Metric: Zung Self-Rating Anxiety Scale (SAS) score (20-80).
Depressive Symptoms | Baseline (T0), End of treatment (T1, after 8 weeks), Follow-up (T2, 4 weeks after end of treatment).
  Changes in depressive symptoms. Metric: Zung Self-Rating Depression Scale (SDS) score (20-80).
Emotional State | Baseline (T0), End of treatment (T1, after 8 weeks), Follow-up (T2, 4 weeks after end of treatment).
  Evaluation of participants' emotional state. Metric: Delighted Terrible Face scale.
Life Satisfaction | Baseline (T0), End of treatment (T1, after 8 weeks), Follow-up (T2, 4 weeks after end of treatment).
  Changes in overall satisfaction with life. Metric: Satisfaction with Life Scale (SWLS) score (5-35).
Positive and Negative Emotions | Baseline (T0), End of treatment (T1, after 8 weeks), Follow-up (T2, 4 weeks after end of treatment).
  Changes in positive and negative affect. Metric: Positive and Negative Affect Schedule (PANAS) scores (10-50 per dimension).
Emotional Regulation Strategies | Baseline (T0), End of treatment (T1, after 8 weeks), Follow-up (T2, 4 weeks after end of treatment).
  Changes in emotional regulation processes, specifically reappraisal and suppression. Metric: Emotional Regulation Questionnaire (ERQ) scores (typical range: 6-42 for Reappraisal, 4-28 for Suppression).

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Paolucci, Associate Professor, MD, PhD, Principal Investigator — University of Study "G. d'Annunzio" of Chieti-Pescara; Ruggero D'Anastasio, Full Professor, Study Director — University of Study "G. d'Annunzio" of Chieti-Pescara, Director of University Museum; Giannapia Affaitati, MD, PhD, Principal Investigator — University of Study "G. d'Annunzio" of Chieti-Pescara, Co-Principal Investigator
Locations (2):
- Italy (2):
  - CARES - Centro per la Disabilità, la Riabilitazione e Medicina dello Sport - University Center, Chieti, Abruzzo
  - Museo Universitario UD'A, Chieti, Abruzzo

IPD SHARING:
Plan to Share IPD: No